CLINICAL TRIAL: NCT07271654
Title: Can Pretreatment With Analgesics Reduce Postendodontic Pain? A Randomized Controlled Trial
Brief Title: Can Pretreatment With Analgesics Reduce Postendodontic Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Faiz ur rahman, Postgraduate Resident, Department of Operative Dentistry, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCD-EndoPain-2025
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Pulpitis - Irreversible
Keywords: Endodontic pain; NSAIDS; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre treatment with NSAIDS (Experimental): Experimental
  Interventions: Procedure: Pre treatment with NSAIDS; Procedure: No pretreatment with NSAIDS.
- No pre treatment with NSAIDS (Active Comparator): No pretreatment medication was administered before endodontic treatment.
  Interventions: Procedure: Pre treatment with NSAIDS; Procedure: No pretreatment with NSAIDS.

INTERVENTIONS:
Procedure: Pre treatment with NSAIDS — Single oral dose of 100 mg Diclofenac Sodium, administered 30 minutes prior to endodontic treatment.
Procedure: No pretreatment with NSAIDS. — Single oral dose of 100 mg Diclofenac Sodium, administered 30 minutes prior to endodontic treatment.

SUMMARY:
This randomized controlled trial investigated whether a single dose of diclofenac sodium taken before a root canal procedure can reduce pain in the hours following the treatment. 160 patients with tooth pain from irreversible pulpitis were divided into two groups. One group received 100mg of diclofenac sodium 30 minutes before their procedure, while the other group received no pretreatment. Pain levels were measured at 6, 12, and 24 hours after the procedure. The study found that patients who took diclofenac before treatment were significantly more likely to be pain-free at 6 and 12 hours after the procedure compared to those who did not.

DETAILED DESCRIPTION:
This was a parallel-arm, randomized controlled trial conducted in the Department of Operative Dentistry, Saidu College of Dentistry. A total of 160 patients aged 20-60 years with a diagnosis of irreversible pulpitis in vital teeth were enrolled via consecutive sampling. Participants were randomized using a computer-generated sequence with allocation concealment via sealed opaque envelopes. The experimental group (n=80) received a single oral dose of 100 mg diclofenac sodium 30 minutes prior to endodontic treatment. The control group (n=80) received no pretreatment medication. All endodontic treatments were performed by experienced operators using a standardized protocol. The primary outcome was postendodontic pain intensity, assessed using a Visual Analogue Scale (VAS) and categorized as none, mild, moderate, or severe. Pain levels were recorded via structured telephone interviews at 6, 12, and 24 hours post-treatment. Statistical analysis was performed using R software, with group comparisons made using the chi-square test.

ELIGIBILITY:
Inclusion Criteria:Pakistani nationals aged 20-60 years. Diagnosis of irreversible pulpitis in a vital tooth (single or multi-rooted), confirmed by a positive cold test.

No evidence of periapical abscess on radiographs. - Exclusion Criteria:Prior use of analgesics within a specified timeframe Presence of periodontal disease.

Current use of prophylactic antibiotics.

Pregnancy or lactation.

Mental disabilities.

Systemic illnesses contraindicating endodontic therapy.

Known hypersensitivity or adverse reaction to NSAIDs.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postendodontic Pain | 6 hours after endodontic treatment
  Proportion of patients reporting no pain, mild pain, moderate pain, or severe pain as measured on a Visual Analogue Scale (VAS

SECONDARY OUTCOMES:
Incidence of Postendodontic Pain | 12 hours after endodontic treatment
  Proportion of patients reporting no pain, mild pain, moderate pain, or severe pain as measured on a Visual Analogue Scale (VAS).
Incidence of Postendodontic Pain | 24 hours after endodontic treatment
  Proportion of patients reporting no pain, mild pain, moderate pain, or severe pain as measured on a Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Saidu College of dentistry,Swat, Swat, Pakistan

IPD SHARING:
Plan to Share IPD: No